CLINICAL TRIAL: NCT01599793
Title: A Phase II Study of MRI Based Functional Imaging for the Evaluation of Bone Metastasis in Men With Castrate Resistant Prostate Cancer Receiving XL184
Brief Title: Magnetic Resonance Imaging in Measuring the Effect of Cabozantinib in Patients With Castrate Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-1031; NCI-2012-00677 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Bone Metastases; Castrate-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer
Keywords: castrate resistant prostate cancer; CRPC; cabozantinib; XL184
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabozantinib; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive cabozantinib PO QD. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cabozantinib; Other: laboratory biomarker analysis; Procedure: magnetic resonance imaging

INTERVENTIONS:
Drug: cabozantinib — Given PO
  Other Names: XL184
Other: laboratory biomarker analysis — Correlative studies
Procedure: magnetic resonance imaging — Undergo MRI
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging

SUMMARY:
This study is being done to help researchers understand more about prostate cancer that has spread to the bones by using the newest magnetic resonance imaging (MRI) techniques and to better understand the effect of an experimental drug called XL184 (or cabozantinib) on bone disease. The other purposes of the study are to better understand the effect of XL184 on prostate cancer progression, bone pain, and on any cancer cells that patients may have circulating within the blood (called circulating tumor cells)

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine effect of XL184 on the functional MRI metrics Ktrans and apparent diffusion coefficient (ADC) within castrate resistant prostate cancer bone metastases.

SECONDARY OBJECTIVES:

I. To quantify progression free survival in men with castrate resistant prostate cancer (CRPC) treated with XL184 according to Prostate Cancer Working Group criteria.

II. To correlate and changes in MRI based functional metrics with bone scan, prostate specific antigen (PSA), Response Evaluation Criteria in Solid Tumors (RECIST) response criteria, circulating tumor cells (CTC) number and with changes in pain.

III. To explore c-MET, phospho-c-MET staining on circulating tumor cells as a predictive biomarker for response and duration of response to XL-184.

OUTLINE:

Patients receive cabozantinib orally (PO) once daily (QD). Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed prostate cancer with progressive disease
* Evidence of castration resistance defined as disease progression despite a testosterone level < 50ng/dL (or surgical castration)
* Evidence of metastatic disease to the bones within the lumbar spine, sacrum, or pelvic bones that is identifiable on screening pelvic MRI
* If patient has had prior pelvis radiation therapy (RT), then bone metastases must be out of radiated port (e.g. lumbar or sacral spine)
* Any prior therapy for castrate disease acceptable other than prior XL184 with a minimum washout of 28 days for any other anticancer therapy
* Patients with castrate resistant disease post antiandrogen therapy/withdrawal must meet at least one of the following criteria:

  * Have not received docetaxel chemotherapy
  * Have received docetaxel chemotherapy but received less then 225mg/m2 cumulative dose
  * Have documented liver metastases
  * Have no pain or pain that does not require a long acting (SR) narcotic
  * Have received mitoxantrone chemotherapy in the past for CRPC

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study
* Patients who are receiving any other investigational agents
* Prior treatment with other vascular endothelial growth factor (VEGF) or c-MET targeted therapies
* History of hematemesis or hemoptysis
* The subject has uncontrolled or significant intercurrent illness
* The patient requires concomitant treatment, in therapeutic doses, with anticoagulants

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-05; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Szmulewitz, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Started | 19
Completed | 17
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 68 [51 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in the Functional MRI Metrics Ktrans Between 2 Weeks and Baseline
Description: Ktrans is a measurement calculating the volume transfer constant of the contrast reagent and essentially is a measurement of vascular perfusion.
  To determine the effect of XL184 on the functional MRI metrics Ktrans, Ktrans parameters were measured at baseline, two week time-point, 12 weeks, and 24 weeks for disease monitoring. Change between baseline and 2 weeks reported.
Time Frame: baseline, 2 weeks
Population: 2 individuals had missing values for Ktrans from baseline to 24 weeks
Measure: Least Squares Mean (Standard Deviation); unit: per minute (or min-1)
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 15
per minute (or min-1) | 0.026 (0.005)
Statistical Analysis 1: Comparison: Treatment (Enzyme Inhibitor Therapy); The least square means of ktrans at different time points (baseline, 2 weeks, 12 weeks, 24 weeks) are estimated by a linear mixed model. Comparison of means at different time points were performed. The primary result reported below is for the difference of means between 2 weeks and baseline; Test type: Equivalence — Testing if the change of ktrans between 2 weeks and baseline = 0 (i.e testing if the difference of means between 2 weeks and baseline =0); p = 0.0016, Mixed Models Analysis

2. Secondary Outcome: Association of Progression Free Survival (PFS) With Ktrans and ADC
Description: Time to progression or progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  The approximate survival after standard therapies in this setting is bleak and in the order of months.
  Too few events for a meaningful statistical analysis; no significant results were obtained in Cox regression analyses.
  Therefore, we calculated the median PFS time and its 95% confidence interval.
Time Frame: From start of treatment to time of progression or death, whichever occurs first, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 17
month | 5.100 [2.900 to 5.700]

3. Secondary Outcome: Changes in Bone Scan Response
Description: Bone Scan Response at weeks 2, 12, and 24 were collected. Change between baseline and 2 weeks are reported Bone Scan Response were measured as increase, decrease, or stable of bone lesions and scored as 1, -1, or 0, respectively, where higher values represent a worse outcome.
Time Frame: baseline, 2 weeks
Population: 6 individual have missing bone lesions data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 11
score on a scale | -0.43750 (0.72744)
Statistical Analysis 1: Comparison: Treatment (Enzyme Inhibitor Therapy); Test type: Other — We calculated Spearman Correlation Coefficient between the percent change in Ktrans (from week 0 to 12) and the bone scan response change. We tested if the coefficient = 0; p = 0.3291, t-test, 2 sided; Spearman Correlation Coefficients = 0.36853

4. Secondary Outcome: Correlation of Percent Change in the Functional MRI Metrics to RECIST Tumor Measurements
Description: The protocol proposed to collect RECIST tumor measurements at weeks 0, 12, and 24.
  However, the data were not collected
Time Frame: baseline, 12 weeks, and 24 weeks
Population: Data on RECIST tumor measurements were not collected
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

5. Secondary Outcome: Change of PSA Between 12 Weeks and Baseline
Description: PSA at weeks 0, 12, and 24 were collected. Change between baseline and 12 weeks are reported
Time Frame: baseline, 12 weeks
Population: At 12 weeks, 4 individual have missing PSA data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 13
ng/mL | 453.04 (998.62)
Statistical Analysis 1: Comparison: Treatment (Enzyme Inhibitor Therapy); Test type: Other — We calculated Spearman Correlation Coefficient between the percent change in Ktrans (from week 0 to 12) and the PSA change. We tested if the coefficient = 0; p = 0.2006, t-test, 2 sided; Spearman Correlation Coefficients = -0.41818

6. Secondary Outcome: Correlation of Percent Change in the Functional MRI Metrics With CTC
Description: The protocol proposed to collect CTC measurements at weeks 0, 12, and 24. However, the data were not collected
Time Frame: baseline, 12 weeks, and 24 weeks
Population: data on CTC were not collected
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in Pain Scale Between 12 Weeks and Baseline
Description: Pain scores are measured at baseline and weeks 12, and 24. Change between baseline and 12 weeks are reported .
  In the pain score ranged from 0 to 10. 10 denotes most pain.
Time Frame: baseline,12 weeks
Population: At 12 weeks, 3 individual have missing pain score data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 14
score on a scale | -1.35714 (3.77455)
Statistical Analysis 1: Comparison: Treatment (Enzyme Inhibitor Therapy); Test type: Other — We calculated Spearman Correlation Coefficient between the percent change in Ktrans (from week 0 to 12) and the Change in pain scale. We tested if the coefficient = 0; p = 0.5828, t-test, 2 sided; Spearman Correlation Coefficients = 0.17669

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed every two weeks for the first three months and then every 4 weeks thereafter (until one year).
Description: Assessment of toxicities and adverse events were graded according to the Common Toxicity Criteria (CTC), version 4.03.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
All-Cause Mortality (participants affected / at risk) | 1/17
Serious Adverse Events (participants affected / at risk) | 4/17
Other Adverse Events (participants affected / at risk) | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=17)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1)
hospitalized with pneumaonia (Aspiration) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Syncope (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=17)
Fatigue (General disorders) | 7 (7)
mucositis (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 2 (2)
plantar erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 2 (2)
elevated transaminases (Gastrointestinal disorders) | 1/1 (1)
decreased appetite (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-08-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT01599793/Prot_SAP_000.pdf